CLINICAL TRIAL: NCT06067178
Title: Effectiveness of a Health Dialogue Intervention Versus Opportunistic Screening in Primary Care for Type 2 Diabetes and Cardiovascular Disease Prevention in Low Socioeconomic Settings - The DETECT Trial
Brief Title: Health Dialogue Intervention Versus Opportunistic Screening for Type 2 Diabetes and Cardiovascular Disease Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NSV22252
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Pragmatic, cluster-randomized trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Dialogue Intervention (Experimental)
  Interventions: Behavioral: Health Dialogue Intervention
- Opportunistic Screening (Experimental)
  Interventions: Other: Opportunistic Screening

INTERVENTIONS:
Behavioral: Health Dialogue Intervention — 1. Lifestyle assessment: All participants fill out a questionnaire to assess behavioral risk factors for CVD and undergo blood tests for cholesterol and blood glucose.
  2. Lifestyle health dialogue: When presenting in person at the primary care center, blood pressure, BMI, and waist-hip ratio will be measured. The results from the questionnaire, blood tests, blood pressure, and body measurements will be summarized using a visual tool, in which risk factors are graded into risk levels to estimate CVD risk. The visual tool will then be used in the health dialogue to discuss risk factors. The health dialogue is conducted by a licensed healthcare professional who has been trained in the methodology. The dialogue will be conducted in a person-centered manner and will aim to motivate and support lifestyle behavior changes when needed. If necessary, medical treatment will be provided according to existing guidelines.
  Arms: Health Dialogue Intervention
Other: Opportunistic Screening — 1. Risk factor assessment: Opportunistic screening entails screening for risk factors (blood pressure, BMI, blood tests for cholesterol and blood glucose, and smoking) among patients visiting the primary care center for another reason. Screening is conducted by a healthcare professional at which the patient has an appointment.
  2. Detected risk factors for CVD are treated according to the existing care programs and guidelines at the primary care center, which should always include lifestyle advice as the first intervention and medication if hypertension is established. In this intervention, there is a more limited assessment of behavioral risk factors; that is, patients are asked about smoking, but assessment of diet, physical activity, or alcohol consumption is not included in the opportunistic screening.
  Arms: Opportunistic Screening

SUMMARY:
Chronic diseases such as cardiovascular disease and diabetes type 2 are major causes of death worldwide. Preventive interventions can be delivered through primary care, as this is the first-line healthcare with which a considerable proportion of the population comes into contact every year. The goal of this cluster-randomized trial is to compare the effects of a Health Dialogue Intervention (HDI) to Opportunistic Screening (OS) in primary care among middle-aged adults with low socioeconomic status. The main questions it aims to answer are:

* What is the short-term change in cardiovascular risk factors, lifestyle behaviors, and perceived quality-of-life among participants offered HDI, as compared to participants offered OS?
* What is the long-term risk of ischemic heart disease, stroke, type 2 diabetes, and death due to cardiovascular disease or type 2 diabetes, among participants offered HDI, as compared to participants offered OS?

DETAILED DESCRIPTION:
DETECT (health Dialogue intErvention versus opporTunistic scrEening in primary Care for Type 2 diabetes and cardiovascular disease prevention) targets the challenges of primary prevention for individuals with low socioeconomic status by implementing and evaluating two preventive interventions, a Health Dialogue Intervention (HDI) and an Opportunistic Screening (OS), conducted in primary care, specifically targeting settings with low socioeconomic status. The interventions will focus on detecting risk factors for CVD and supporting changes in unhealthy lifestyle behaviors.

The study is designed as a parallel cluster-randomized trial with two conditions, with primary care centers (PCCs) serving as the unit of randomization and individual patients as units of observation for primary and secondary outcomes. Participants randomized to the HDI intervention will be invited to partake in a systematic screening of cardiovascular and metabolic risk factors using questionnaires, blood sampling, and clinical examinations, all of which together form the risk profile. Next, they will be invited to an individually oriented health dialogue which is prescribed by a care provider. The dialogue focuses on promoting healthy lifestyle behaviors and is based on the screening results and the given risk profile. The effects of HDI will be compared to that from OS, wherein participants will be recruited upon scheduling of an appointment at their PCC for any reason, except for individuals with pre-scheduled appointments related to hypertension, T2D, and CVD. Participants receiving OS will be screened for hypertension, overweight/obesity, tobacco usage, blood-lipid profile, and blood glucose.

Short-term outcomes will be assessed at baseline, and 6 and 12-months after receiving the intervention, and long-term outcomes (i.e. 5 and 10 years post intervention) using nationwide registers.

The goal is to recruit a total of 30 PCCs (n=15 in each arm) in the county of Stockholm. Based on real observed variance in levels of systolic blood pressure in the county of Stockholm and accounting for clustering effects, the investigators calculate that a minimum of 840 participants (n=420 in each arm and n=28 per cluster) would yield 80% power to detect a reduction of 5 mmHg systolic blood pressure in the HDI group. To allow for the expected difficulties with recruitment and subsequent attrition, the investigators therefore aim to recruit n=100 patients per cluster, yielding a total study population of 3000.

The core tool of analysis will be a hierarchical model consisting of two levels, individuals and PCCs. The primary model for analyzing changes in systolic blood pressure (primary outcome), other risk factors, lifestyle behaviors, and quality-of-life over 6 and 12 months, will be a mixed-effects Generalized Linear Model to capture variability between and within PCCs. In these models, the treatment effect (HDI versus OS) will be assessed using a fixed effect represented by a dummy variable at PCC level, specifying the type of treatment (HDI/OS). Together, this enables the estimation of the average treatment effect, while accounting for the hierarchical structure of the data. We will estimate unadjusted effects and effects adjusted both/either at the individual level and PCC level, e.g., adjusted for demographic characteristics, socioeconomic status, CNI level, and baseline values of the referred outcome. The analysis will be conducted on an intention-to-treat basis. Potential effect modification will be explored through subgroup analyses and interaction analyses considering sex, birth country, and socioeconomic characteristics. A sensitivity analysis will be conducted to assess whether the individual randomization of a single PCC introduced bias. Thus, we will perform analyzes both including and excluding this PCC.

For the assessment of T2D and CVD incidence and mortality during the extended 5 and 10 years of follow-up, we will calculate hazard ratios using a mixed-effect Cox regression. We will also calculate the number needed to treat (NNT) as 1/absolute risk reduction.

Finally, we also aim to estimate the time needed to treat (TNT) for the interventions. The TNT is a new method designed to consider clinician's time as a finite resource, with the aim of facilitating for guideline committees who develop clinical practice guidelines. The TNT can be expressed in three different ways: 1) the clinician time needed to improve the outcome for one person (TNTNNT), 2) the clinician time needed to provide the intervention for all eligible in a population (absolute TNT), 3) the proportion of the total clinician time available for patient care needed to implement the intervention for everyone eligible (relative TNT). More detailed information on the TNT method and its assumptions is available elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Primary care centres with a Care Need Index above 1.0
* Patients listed at the participating primary care centers.

Exclusion Criteria:

• None.

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure (mmHg) | Baseline (defined as time of HDI/OS), 6 months post intervention, 12 months post intervention
  Measured by care providers in accordance with routine guidelines

OTHER OUTCOMES:
Change in blood cholesterol levels | Baseline, 6 months post intervention, 12 months post intervention
  Measured by care providers in accordance with routine guidelines
Change in blood glucose levels | Baseline, 6 months post intervention, 12 months post intervention
  Measured by care providers in accordance with routine guidelines
Change in body-mass-index | Baseline, 6 months post intervention, 12 months post intervention
  Measured by care providers in accordance with routine guidelines
Change in quality-of-life | Baseline, 6 months post intervention, 12 months post intervention
  Measured by EQ-5D (EuroQol-5 Dimension). From the five dimensions, a summary index is derived, with a maximum score of 1, where 1 indicates the best health state.
Change in tobacco usage | Baseline, 6 months post intervention, 12 months post intervention
  Measured by self-reported questionnaires
Change in dietary habits | Baseline, 6 months post intervention, 12 months post intervention
  Measured by self-reported questionnaires
Change in alcohol consumption | Baseline, 6 months post intervention, 12 months post intervention
  Measured by self-reported questionnaires
Change in physical activity | Baseline, 6 months post intervention, 12 months post intervention
  Measured by self-reported questionnaires
Incidence of ischemic heart disease | 5 and 10 years post intervention
  Collected from national registries
Incidence of stroke | 5 and 10 years post intervention
  Collected from national registries
Incidence of type 2 diabetes | 5 and 10 years post intervention
  Collected from national registries
Mortality due to cardiovascular disease or type 2 diabetes | 5 and 10 years post intervention
  Collected from national registries
Healthcare costs in the health dialogue group vs. the opportunistic screening group | 12 months post intervention
  Administrative data collected form health care providers
Costs per attained blood pressure target among individuals in the health dialogue group vs. the opportunistic screening group | 12 month post intervention
  Administrative data collected form health care providers

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Augustsson, PhD, Principal Investigator — Center for epidemiology and community medicine, Region Stockholm
Locations (1):
- Center for epidemiology and community medicine, Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in accordance with Swedish law and regulations.

REFERENCES:
- [Derived] Ballin M, Backman Enelius M, Dini S, Galanti MR, Hagstromer M, Heintz E, Lager A, de Leon AP, Lundh L, Nystrand C, Walldin C, Augustsson H. Health dialogue intervention versus opportunistic screening in primary care for type 2 diabetes and cardiovascular disease prevention in settings with low socioeconomic status (DETECT): study protocol for a pragmatic cluster-randomized trial. Trials. 2024 Oct 12;25(1):672. doi: 10.1186/s13063-024-08533-8. PMID 39394167